CLINICAL TRIAL: NCT03419702
Title: Effects of Almond Consumption on Chronic Glucose Regulation, Vascular Function and Cognitive Performance: The AL-INCLUSIVE Trial
Brief Title: Almonds and Health Effects on Metabolism, Vascular Function and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: METC173015
Record Dates: First submitted 2018-01-09; First posted 2018-02-05 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: PreDiabetes; Impaired Glucose Tolerance; Impaired Fasting Glucose; Overweight and Obesity
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No almonds
- Experimental (Experimental): Almonds
  Interventions: Dietary Supplement: Almonds

INTERVENTIONS:
Dietary Supplement: Almonds — During the intervention period of 5 months, subjects will receive daily 50 gr almonds. Subjects are free to consume the almonds during the day whenever they want to, i.e. there will not be guidelines when to consume the almonds.
  Arms: Experimental

SUMMARY:
The primary objective of the proposed study is to examine and understand the impact of long-term almond consumption on chronic glucose metabolism in subjects with impaired glucose tolerance and/or impaired fasting glucose.

DETAILED DESCRIPTION:
Objectives:

Secondary objectives are to investigate if improved chronic glucose metabolism in subjects with impaired glucose tolerance and/or impaired fasting glucose after long-term almond consumption translates into improved peripheral and brain vascular function, and enhanced cognitive performance. In addition, the investigators will address to what extent improved chronic glucose metabolism in subjects with impaired glucose tolerance and/or impaired fasting glucose after long-term almond consumption can be explained by (combined) effects of lowered hepatic lipid accumulation and inflammation, skeletal muscle characteristics, visceral and subcutaneous fat accumulation, pancreatic function or fecal microbiota composition.

Study design:

The proposed study will be a 12 months randomised, controlled trial with a cross-over design. Two experimental periods of five months will be separated by a two months washout period.

Study population:

Forty-three impaired glucose tolerant and/or impaired fasting glucose subjects, with overweight and mild obesity (BMI 25-35 kg/m2), aged 40-70 years.

Intervention:

During the intervention period of 5 months, subjects will receive daily 50 gr almonds, but not in the 2 months washout and 5 months control periods.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40-70 years
* Men and women
* BMI between 25-35 kg/m2 (overweight and obese)
* Being classified as having impaired glucose tolerance (IGT) and/or impaired fasting glucose (IFG). IGT is defined according the criteria of the WHO and American Diabetes Association (ADA) as two-hour glucose concentrations of 7.8 to 11.0 mmol/l (140 to 199 mg per dL) during the 75-g oral glucose tolerance test. IFG is defined as having a fasting plasma glucose between 6.1 and 7.0 mmol/l (110 to 125 mg per dL) and a two-hour glucose concentration below 7.8 mmol/l (140 mg per dL).
* Serum total cholesterol < 8.0 mmol/L (further testing is recommended for excessive hyperlipidemia [serum total cholesterol ≥ 8.0 mmol/L] according to the Standard for cardiovascular risk management of the Dutch general practitioners community [NHG])
* Serum triacylglycerol < 4.52 mmol/L
* No current smoker
* No diabetic patients
* No familial hypercholesterolemia
* No abuse of drugs
* Not more than 4 alcoholic consumption per day with a maximum of 21 per week
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* No use of medication known to treat blood pressure, lipid or glucose metabolism
* No use of an investigational product within another biomedical intervention trial within the previous 1-month
* No severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* No active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit
* Willing to comply to study protocol during study
* Informed consent signed

Exclusion Criteria:

* Allergy or intolerance to almonds
* Serum total cholesterol ≥ 8.0 mmol/L
* Serum triacylglycerol ≥ 4.52 mmol/L
* Current smoker, or smoking cessation <12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 4 alcoholic consumptions per day or 21 per week
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Use medication known to treat blood pressure, lipid or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Not willing to give up being a blood donor from 8 weeks before the start of the study, during the study or for 4 weeks after completion of the study
* Not or difficult to venipuncture as evidenced during the screening visit
* Use of over-the-counter and prescribed medication or supplements, which may interfere with study measurements to be judged by the principal investigator;
* Use of oral antibiotics in 40 days or less prior to the start of the study;
* Blood donation in the past 3 months before the start of the study
* Not willing to comply to study protocol during study or sign informed consent

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Change from control period (week 22 and week 52)
  Glucose infusion rate during a hyper-insulinemic euglycemic clamp.

SECONDARY OUTCOMES:
Glucose concentrations | Glucose will be measured at week 0, week 5, week 10, week 21, week 22, week 30, week 35, week 40, week 51, week 52
  Fasting plasma glucose concentrations will be determined in blood samples.
Markers for fasting lipid metabolism | These markers will be measured at week 0, week 5, week 10, week 21, week 22, week 30, week 35, week 40, week 51, week 52
  Markers for fasting lipid metabolism include serum total cholesterol (mmol/L), HDL cholesterol (mmol/L), and triacylglycerol (mmol/L) concentrations.
LDL cholesterol concentrations | These markers will be calculated from measurements at week 0, week 5, week 10, week 21, week 22, week 30, week 35, week 40, week 51, week 52
  Fasting LDL cholesterol concentrations will be determined in blood samples using the Friedewald equation.
C-reactive protein concentrations | CRP will be measured at week 0, week 5, week 10, week 21, week 22, week 30, week 35, week 40, week 51, week 52
  Concentrations of CRP will be determined in blood samples.
Blood pressure | Blood pressure will be measured at week 0, week 5, week 10, week 21, week 22, week 30, week 35, week 40, week 51, week 52
  Systolic and diastolic blood pressure.
Body weight | Body weight will be measured at week 0, week 5, week 10, week 21, week 22, week 30, week 35, week 40, week 51, week 52
  Body weight in kg.
Body circumferences | Waist and hip circumferences will be measured at week 0, week 5, week 10, week 21, week 22, week 30, week 35, week 40, week 51, week 52
  Waist and hip circumferences.
Pulse Wave Analysis | Change from control period (week 21 and week 51)
  Vascular function (arterial stiffness).
Pulse Wave Velocity | Change from control period (week 21 and week 51)
  Vascular function (arterial stiffness).
Retinal microvascular caliber | Change from control period (week 21 and week 51)
  Arteriovenous ratio and diameter of retinal arterioles and venules will be measured by retinal microvascular imaging.
Cognitive performance | Cognition will be tested at week 0, week 10, week 21, week 30, week 40, week 51.
  Cambridge Neuropsychological Test Automated Battery.
Markers for low-grade systemic inflammation | Change from control period (week 21 and week 51)
  Markers for low-grade systemic inflammation include IL-6, IL-8, TNF-alpha and SAA.
Markers for endothelial dysfunction | Change from control period (week 21 and week 51)
  Markers for endothelial dysfunction include sVCAM-1, sICAM-1 and soluble E-selectin.
Markers for postprandial lipid metabolism | Change from control period (week 21 and week 51)
  Markers for postprandial lipid metabolism include triacylglycerol (mmol/L) and NEFA concentrations.
Markers for fasting and postprandial glucose and insulin metabolism | Change from control period (week 21 and week 51)
  Markers for fasting and postprandial glucose and insulin metabolism include plasma glucose, serum insulin, C-peptide and HbA1c concentrations. Also HOMA-IR will be calculated.
Markers for liver function | Change from control period (week 21 and week 51)
  Markers for liver function include ALAT and ASAT concentrations.
Markers for nerve growth | Change from control period (week 21 and week 51)
  Markers for nerve growth include BDNF concentrations.
Markers for advanced glycation endproducts | Change from control period (week 21 and week 51)
  Markers for advanced glycation endproducts include dicarbonyl, CML, CEL and MG-H1 concentrations.
Nitric oxides concentrations | Change from control period (week 21 and week 51)
  Concentrations of NOx will be determined in blood samples.
Cerebral blood flow | Change from control period (week 22 and week 52)
  Arterial Spin labeling will be performed to determine cerebral blood flow.
Fat distribution in abdomen | Change from control period (week 22 and week 52)
  Magnetic Resonance Imaging measurements will be included to quantify abdominal fat compartments (i.e. subcutaneous and visceral fat) and fat content of abdominal organs (i.e. liver and pancreas).
Biopsies adipose tissue | Change from control period (week 22 and week 52)
  Fat biopsies to examine fat cell size and inflammation in adipose tissue.
Biopsies muscle tissue | Change from control period (week 22 and week 52)
  Muscle biopsies to examine mitochondrial function.
Lipid oxidation | Indirect calorimetry will be performed at week 21, week 22, week 51, week 52 at several time slots.
  Energy expenditure and substrate metabolism will be calculated from measurements via indirect calorimetry during the postprandial test.
Glucose oxidation | Indirect calorimetry will be performed at week 21, week 22, week 51, week 52 at several time slots.
  Energy expenditure and substrate metabolism will be calculated from measurements via indirect calorimetry during the postprandial test.
Blood pressure profiles | Change from control period (week 21 and week 51)
  Blood pressure profiles will be measured for 48 hr via a Mobil-O-Graph.
Glucose profiles | Change from control period (week 21 and week 51)
  Glucose profiles will be measured for 48 hr using the FreeStyle Libre Pro.
Physical activity profiles | Change from control period (week 21 and week 51)
  Physical activity patterns will be monitored for 48 hr with the MOX device.
Microbiota composition | Change from control period (week 21 and week 51)
  Fecal samples to be used for analysing microbiota composition will be collected.
General well-being | General well-being will be tested at week 0, week 10, week 21, week 30, week 40, week 51.
  Quality of life and Affect grid questionnaires will be assessed.
Food frequency | Food frequency will be tested at week 0, week 10, week 21, week 30, week 40, week 51.
  Food frequency questionnaire will be assessed.
Skinfold measurements | Change from control period (week 22 and week 52)
  Calliper testing for determining body fat composition.

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, PhD, Principal Investigator — Maastricht University; Ronald P Mensink, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Department of Nutrition and Movement Sciences, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chavez-Alfaro MA, Mensink RP, Gravesteijn E, Joris PJ, Plat J. Effects of long-term almond consumption on markers for vascular function and cardiometabolic risk in men and women with prediabetes: results of a randomized, controlled cross-over trial. Eur J Nutr. 2024 Nov 15;64(1):7. doi: 10.1007/s00394-024-03510-y. PMID 39546040
- [Derived] Gravesteijn E, Mensink RP, Plat J. The effects of long-term almond consumption on whole-body insulin sensitivity, postprandial glucose responses, and 48 h continuous glucose concentrations in males and females with prediabetes: a randomized controlled trial. Eur J Nutr. 2023 Sep;62(6):2661-2672. doi: 10.1007/s00394-023-03178-w. Epub 2023 May 31. PMID 37258943